CLINICAL TRIAL: NCT05876689
Title: Swept Source OCT Imaging With the DREAM VG-OCT
Status: Completed | Type: Observational
Sponsor: Robert T. Chang, MD (Other)
Responsible Party: Sponsor-Investigator, Robert T. Chang, MD, Associate Professor of Ophthalmology, Stanford University
Organization: Stanford University (Other)
Other Study IDs: 70411
Record Dates: First submitted 2023-05-17; First posted 2023-05-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Eye Diseases; Myopia; Glaucoma
MeSH Terms: conditions — Eye Diseases; Myopia; Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- DREAM OCT: All 50 patients will have both eyes (if able) imaged, 3 times, on the same day during their clinic visit.
  Interventions: Device: DREAM OCT

INTERVENTIONS:
Device: DREAM OCT — Swept Source OCT (similar to Zeiss Plex Elite)

SUMMARY:
The Intalight Dream OCT is the first combo anterior plus posterior device to perform both OCT and OCT-A at depth of 16mm. This is especially useful in patient who are very nearsighted as it allows us to image all in one frame. The intention of this study is to see how the images differ on the same patients when compared to the Cirrus OCT and to test for the repeatability of the images on a single day.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18
* Myopes with a current or previously documented spherical equivalent refraction < -4D
* At least half of the subjects should have had at least one Cirrus OCT RNFL and macula performed as well as a Humphrey visual field performed in those with OCT abnormalities

Exclusion Criteria:

* Unable to comply with study imaging
* unclear ocular media
* Participant has, in the opinion of the investigator, any physical or mental condition that would affect the participation in the study or may interfere with the study procedures, evaluations and outcome assessments.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The investigators will be imaging 100 eyes (50 patients unless there are monocular patients) from all genders and ethnic backgrounds who are moderate-high myopes with or without the diagnosis of glaucoma.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Assessing difference in intraocular structures | Baseline
  Assessing the performance of the DREAM VG OCT scan patterns in high myopes including glaucomatous eyes to see if there are differences in the lamina cribrosa structure when compared to patients previous Cirrus OCTs.
Assessing difference in intraocular vascular structures | Baseline
  Assessing differences in vascular density in areas with presumed myopic-related field defects vs. low tension glaucoma perimetric disease

SECONDARY OUTCOMES:
Assessing repeatability of scans | Baseline
  Analyze the repeatability of quantitative RNFL and GCC parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Chang, MD, Principal Investigator — Stanford University
Locations (1):
- Byers Eye Institute, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No